CLINICAL TRIAL: NCT07245420
Title: Evaluation Of Cardiovascular Health Outcomes Among Survivors 2 (ECHOS2)
Brief Title: Evaluation Of Cardiovascular Health Outcomes Among Survivors 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ECHOS2; 1R01CA297448 (NIH); NCI-2025-07891 (Other: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2025-11-03; First posted 2025-11-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Health Behavior
Keywords: Childhood Cancer Survivors; Cardiomyopathy Screening; eHealth Intervention
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (Active Comparator): Participants receive a personalized survivorship care plan and educational materials about cardiomyopathy risk and screening recommendations.
  Interventions: Behavioral: Survivorship Care Plan + Educational Materials (delivered via CIAS platform)
- Healthy Hearts eHealth Intervention (Experimental): Participants receive the same SOC materials plus a tailored eHealth intervention using CIAS. This includes avatar-led motivational interviewing, survivor video vignettes, and interactive modules addressing screening barriers.
  Interventions: Behavioral: Healthy Hearts eHealth Program

INTERVENTIONS:
Behavioral: Survivorship Care Plan + Educational Materials (delivered via CIAS platform) — Participants receive a personalized survivorship care plan and educational materials about cardiomyopathy risk and screening recommendations. Materials are delivered via the CIAS platform and include infographics, treatment summaries, and general information about screening.
  Arms: Standard of Care (SOC)
Behavioral: Healthy Hearts eHealth Program — Participants receive the same SOC materials plus a tailored, interactive eHealth intervention delivered via the CIAS platform. This includes avatar-led motivational interviewing (MI), survivor video vignettes, interactive modules addressing perceived barriers, self-efficacy, and goal setting. The intervention is designed to mimic MI counseling in a scalable format.
  Arms: Healthy Hearts eHealth Intervention

SUMMARY:
Childhood cancer survivors who received certain treatments are at a higher risk of developing heart problems in the future. This study is looking at ways to educate childhood cancer survivors about that risk and encourage them to receive a recommended heart screening test.

DETAILED DESCRIPTION:
Primary Objective:

* To determine the efficacy of the Healthy Hearts eHealth intervention compared to standard of care for improving screening echocardiogram adherence in childhood cancer survivors.

Secondary Objective

* To determine the efficacy of the Healthy Hearts eHealth intervention compared to standard of care for improving mediators of screening echocardiogram adherence in childhood cancer survivors.

After consenting, participants will complete a survey that will take about 15-20 minutes to complete. After this survey, they will be randomly assigned to participate in the Healthy Hearts eHealth Intervention or to receive standard educational materials about hearth health screening.

All participants will receive the Standard of Care (SOC) materials delivered via the Computerized Intervention Authoring System (CIAS) platform (i.e., a personalized survivorship care plan and educational materials regarding cardiomyopathy risk and need for screening). In addition to the SOC materials received by controls, the Healthy Hearts eHealth intervention arm will receive CIAS platform delivered Motivational Interview (MI), including scripted interaction with an avatar, video vignettes, and patient testimonials

ELIGIBILITY:
Inclusion Criteria:

* Childhood Cancer Survivor Study (CCSS) Participants
* Age ≥26 years
* Treated with cumulative doxorubicin equivalent anthracycline doses ≥100 mg/m2 with any/no radiation, or ≥15 Gy chest radiation with any/no anthracyclines
* No history of cardiomyopathy
* Has not had an echocardiogram in the previous 5 years
* Has a history of successful completion of CCSS surveys
* English-Speaking
* Has not been enrolled in ECHOS-1 (pilot)

Exclusion Criteria:

• Currently participating in a long-term follow-up program that provides risk-based screening

Min Age: 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Received Cardiomyopathy Screening at 12 months between Participants Randomized to the Healthy Hearts eHealth Intervention group as compared to the standard of care. | 12 months
  This outcome will be measured through self-reported questionnaire at 12 months along with confirmation through medical record review.
Difference in Precursors to Cardiomyopathy Screening at 12 months between Participants Randomized to the Healthy Hearts eHealth Intervention group as Compared to the Standard of Care. | 12 months
  This outcome will use questions included in the baseline and 12 month questionnaire to calculate the differences in precursors to cardiomyopathy screening (perceived barriers, knowledge, motivation, beliefs, self-efficacy) at 12 months between participants randomized to Healthy Hearts eHealth Intervention vs participants assigned to standard care.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Ehrhardt, MD, MS, MPI, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols